CLINICAL TRIAL: NCT04529642
Title: Is the 6-Minute Walking Test Combined With an IMU Useful in Stroke Rehabilitation Assessment? A Pilot Observational Study
Brief Title: Is the 6-Minute Walking Test Combined With an IMU Useful in Stroke Rehabilitation Assessment?
Status: Completed | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Other Study IDs: JP-001
Record Dates: First submitted 2020-08-11; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Stroke; Physical Therapy Modalities; Gait Analysis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke Group: Inclusion criteria were as follows: age above 18, Mini-Mental State Examination ≥ 24, ability to provide written informed consent and to understand the test instructions, and the presence of a single stroke. Exclusion criteria were as follows: more than one stroke, stroke area other than the cerebral cortex, or concomitant neurological disease and pathology of the locomotor system. This group has been analysed also dividing the subjects according to the stroke phase in 3 subgroups: Acute phase group, Subacute phase group, Chronic stroke group
  Interventions: Diagnostic Test: Inertial Measurement Unit evaluation
- Healthy Group: Healthy subjects age matched with the stroke group
  Interventions: Diagnostic Test: Inertial Measurement Unit evaluation

INTERVENTIONS:
Diagnostic Test: Inertial Measurement Unit evaluation — An IMU was worn by the subjects during the execution of the 6MWT, to assess the kinematic parameters of gait.

SUMMARY:
This Observational study aims at the evaluation of stroke subjects with an inertial measurement unit (IMU) during the execution of a 6-Minute Walking test, to evaluate the associations between the kinematic parameters retrieved trough an IMU and the classical outcome scales. Moreover compare the stroke subjects with age-matched healthy subjects, and detect the differences of gait kinematic.

ELIGIBILITY:
Stroke Group

Inclusion Criteria:

* Age >= 18;
* Mini-Mental State Examination ≥ 24;
* Ability to provide written informed consent and to understand the test instructions;
* Presence of a single stroke.

Exclusion Criteria:

* More than one stroke;

  . Stroke area other than the cerebral cortex;
* Concomitant neurological disease and pathology of the locomotor system.

Healthy Group

Inclusion Criteria:

- Volunteers with age similar to the Stroke group subjects

Exclusion Criteria:

- Any disease that could affect the performance in terms of metres walked and quality of gait.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stroke Group:
  Post stroke subjects who were referred to the centre for rehabilitation, and were able to independently walk with or without an assistive device.
  Healthy Group:
  Healthy controls age-matched with the subjects in the stroke group
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Temporal parameters of gait | 1 day
  Assessed through an Inertial Measurement Unit, it include the time length of steps, of the stance phase, of double and single limb support phase.
Canadian Neurological Stroke Scale | Baseline
  To state the stroke condition
Berg Balance Scale | Baseline
  To assess the balance of stroke subjects
Motricity Index | Baseline
  To assess the strength of stroke subjects
Gait speed | 1 day
  Assessed through an Inertial Measurement Unit, in different moments of the 6-Minute walking test.
Meters walked | 1 day
  The amount of meters walked in 6 minutes
Step Cadence | 1 day
  Amount of steps for each minute
Symmetry | 1 day
  AN index of the symmetry between the two sides of the subjects during gait

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided